CLINICAL TRIAL: NCT06222138
Title: Study of Biologic Tumor and Plasma Biomarkers of Response to TTFields in Patients Treated for Newly Diagnosed Glioblastoma
Acronym: EXOFIELDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23 TETE 04
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Biologic tumor and plasma biomarkers; Translational research; TTFields
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with newly diagnosed glioblastoma (Experimental)
  Interventions: Other: The samples described below will be collected:

INTERVENTIONS:
Other: The samples described below will be collected: — For each included patient, blood samples will be collected during baseline visit (before initiation of radio-chemotherapy), then before initiation of TTFields and every 3 months during TTFields treatment. Additional blood samples will be scheduled at recurrence (if applicable).
  Moreover, tumor samples (formalin paraffin embedded (FFPE) tumor block and fresh samples) will be collected from surgery specimen on primary tumor by the sponsor for analysis. In case of recurrence, and if a second surgery is possible, tumor samples will also be collected.
  Tumor samples will be collected from biopsies taken in the course of routine practice and from surgical specimens collected during surgical procedure.

SUMMARY:
This trial is a translational, open-label, monocentric prospective study of 80 patients aiming to study resistance mechanisms as well as biomarkers of resistance or sensitivity to TTFields.

The study will be conducted on a population of patients with newly diagnosed glioblastoma treated with radio-chemotherapy followed by TTFields in the context of either routine care or a clinical trial.

In this study, the Optune® system (battery operated device which delivers TTFields to the brain) will not be under investigation.

For each included patient, blood samples will be collected during baseline visit (before initiation of radio-chemotherapy), then before initiation of TTFields and every 3 months during TTFields treatment. Additional blood samples will be scheduled at recurrence (if applicable).

Moreover, tumor samples (formalin paraffin embedded (FFPE) tumor block and fresh samples) will be collected from surgery specimen on primary tumor by the sponsor for analysis. In case of recurrence, and if a second surgery is possible, tumor samples will also be collected.

Tumor samples will be collected from biopsies taken in the course of routine practice and from surgical specimens collected during surgical procedure. No additional biopsies will be performed for the study.

Patients will be followed-up for time to progression and overall survival for a maximum duration of 24 months from the TTFields initiation.

MRI performed by patients during the course of the study will be collected by the sponsor for additional future research purposes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of study entry.
2. Patient with newly diagnosed glioblastoma.
3. Patient for which a treatment with radio-chemotherapy followed by TTFields has been decided and has not been started.
4. Signed written informed consent.
5. Patient able to participate and willing to give informed consent prior performance of any study-related procedures and to comply with the study protocol
6. Patient affiliated to a Social Health Insurance in France.

Exclusion Criteria:

1. Any condition contraindicated with sampling procedures required by the protocol.
2. Any contraindication to the use of the medical device administering TTFields.
3. Simultaneous participation in a therapeutic interventional clinical trial.
4. Patient pregnant, or breast-feeding.
5. Known history of positive test for hepatitis B virus or hepatitis C virus or human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
6. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure
7. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) defined as the time from inclusion until death from any cause or last follow-up (censored data). | 27 months for each patient
Time to Progression (TTP) defined as the time from inclusion until progression. Patients without progression are censored at last follow-up. | 27 months for each patient

SECONDARY OUTCOMES:
Number of patients with MRI collected. | 27 months for each patient

CONTACTS AND LOCATIONS:
Locations (1):
- IUCT-O, Toulouse, France